CLINICAL TRIAL: NCT03820505
Title: Observatory of Unintentional Births Hospital Extras in Hérault
Brief Title: Observatory of Unintentional Births Hospital Extras
Acronym: AIEH34
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: SDIS34 - MONTPELLIER (Unknown); SAMU CHU Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0442
Record Dates: First submitted 2019-01-23; First posted 2019-01-29 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Unexpected Delivery Outside Maternity
Keywords: obstetrics; pre-hospital emergencies unannounced delivery outside maternity,; mortality-morbidity; reinforcement midwife in pre-hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, pre-hospital unexpected birth is a rare situation, but over the last ten years, the investigators have seen an increase in the number of these.

For this, the investigators realize an observatory of these deliveries and their care from the call for help and the investigators continue the follow-up and the future of patients and newborns until J7 postpartum.

DETAILED DESCRIPTION:
As a result, the investigators also found a very high variability in the number of deliveries per month for the EMS 34 and the SSSM of the SDIS 34, which can reach up to 11 deliveries per month (May 2014 example).

Formalized expert recommendations were published in 2010 by SFAR, which then led to the establishment of a national observatory for IEA at the end of 2011, in which the investigators have been participating for 4 years.

Currently the national database lists 2000 unannounced deliveries including 230 in the Hérault.

This observational study allows us to evaluate the management of these patients and newborns, the risks and needs of pre-hospital teams, including the need for reinforcement and expertise of midwives.

The investigators can also assess mortality and morbidity, as well as the extension of hospital stays beyond J7

ELIGIBILITY:
Inclusion Criteria:

* Unexpected delivery outside maternity, presence of a medical team during the care

Exclusion Criteria:

* Absence of medicalization

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Unexpected delivery outside maternity in the Hérault department
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
number of unexpected hospital deliveries (AIE) | DAY 0 TO DAY 7 TO DELIVRERY
  Estimate the impact of non-maternal AIE by the SMUR and the SSM in the department of Héraul, and compare it to the national overall activity

SECONDARY OUTCOMES:
Method of taking care of unannounced extra hospital deliveries | DAY 0 TO DAY 7 POST DELIVRERY
  Method of taking care of unannounced extra hospital deliveries
Difficulties during an unexpected delivery outside maternity | DAY 0 TO DAY 7 POST DELIVRERY
  Identify the difficulties during an unexpected delivery outside maternity
Risks during an unexpected delivery outside maternity | DAY 0 TO DAY 7 POST DELIVRERY
  Identify the risks during an unexpected delivery outside maternity
Possible immediate complications during an unexpected delivery outside maternity | DAY 0 TO DAY 7 POST DELIVRERY
  Identify the possible immediate complications during an unexpected delivery outside maternity

CONTACTS AND LOCATIONS:
Overall Officials: Christelle GRAF, wise woman, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC